CLINICAL TRIAL: NCT01319409
Title: Single- vs. Double-Bundle ACL Reconstruction: A Prospective Randomized Trial
Brief Title: Single- vs. Double-Bundle ACL Reconstruction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO09020493; R01AR056630-01A2 (NIH)
Record Dates: First submitted 2011-03-15; First posted 2011-03-21 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: Anterior cruciate ligament surgery; Anterior cruciate ligament reconstruction; Single bundle anterior cruciate ligament reconstruction; Double bundle anterior cruciate ligament reconstruction; Randomized clinical trial
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anatomic Double-Bundle ACL Reconstruction (Experimental): Subjects in this arm will undergo anatomic double-bundle ACL reconstruction using an autograft quadriceps tendon with a bone block. The graft will be split into 2 strands, 1 to recreate the posterolateral (PL) bundle, the other to recreate the anteromedial (AM) bundle of the ACL. The bone block will be placed in a single femoral tunnel located in the center of the femoral ACL insertion site. The free ends of the graft will be placed in tunnels located in the centers of the tibial insertions for the PL and AM bundles. The PL bundle will be fixed with the knee in full extension and the AM bundle will be fixed with the knee at 45 degrees of flexion.
  Interventions: Procedure: Anatomic Double-Bundle ACL Reconstruction
- Anatomic Single-Bundle ACL Reconstruction (Active Comparator): Subjects in this arm will undergo anatomic single-bundle ACL reconstruction using an autograft quadriceps tendon with a bone block. The graft will not be split. The bone block will be placed in a single femoral tunnel located in the center of the femoral ACL insertion site. The free end of the graft will be placed in single tunnel located in the center of the tibial ACL insertion site. The graft will be fixed with the knee at 10 20 20 degrees of flexion.
  Interventions: Procedure: Anatomic Single-Bundle ACL Reconstruction

INTERVENTIONS:
Procedure: Anatomic Double-Bundle ACL Reconstruction — Surgical reconstruction of the posterolateral (PL) and anteromedial (AM) bundles of the ACL using an autograft quadriceps tendon with a bone block that is split into 2 free arms to recreate the AM and PL bundles. The bone block is placed in a single femoral tunnel located in the center of the femoral ACL insertion site. The free ends of the graft are be placed in 2 separate tunnels located in the centers of the tibial insertions for the PL and AM bundles. The PL bundle is fixed with the knee in full extension and the AM bundle is fixed with the knee at 45 degrees of flexion.
  Arms: Anatomic Double-Bundle ACL Reconstruction
Procedure: Anatomic Single-Bundle ACL Reconstruction — Surgical reconstruction of the ACL using a single autograft quadriceps tendon with a bone block. The free end of the graft is not split. The bone block is placed in a single femoral tunnel located in the center of the femoral ACL insertion site. The single free end of the graft is placed in a single tibial tunnel located in the center of the tibial ACL insertion site. The graft is fixed with the knee in 10 to 20 degrees of flexion.
  Arms: Anatomic Single-Bundle ACL Reconstruction

SUMMARY:
The purpose of this double-blind, randomized clinical trial to compare outcomes of single-bundle (SB) to anatomic double-bundle (DB) ACL reconstruction. We hypothesize that anatomically reconstructing both bundles of the ACL will lead to better restoration of healthy knee mechanics and clinical outcomes. In addition to standard clinical outcome measures, we will utilize a unique combination of high-speed biplane radiography (for highly accurate assessment of knee kinematics) and 3D imaging (MRI and CT, to define joint and cartilage morphology) to characterize joint kinematics and cartilage surface interactions during functional tasks.

The specific aims of this study are to:

Specific Aim 1: Determine if anatomic double-bundle ACL reconstruction restores normal dynamic knee function better than single-bundle ACL reconstruction.

Hypothesis 1.1 Knee kinematics after anatomic double-bundle ACL reconstruction are more similar to the uninjured contra-lateral limb than after single-bundle ACL reconstruction, as measured with dynamic stereoradiography 6 and 24 months after surgery.

Hypothesis 1.2 Graft elongation from 6 to 24 months after surgery is reduced with anatomic double-bundle ACL reconstruction in comparison to single-bundle ACL reconstruction, as measured with dynamic stereoradiography.

Specific Aim 2: Determine if anatomic double-bundle ACL reconstruction results in better clinical outcomes than single-bundle ACL reconstruction.

Hypothesis 2.1 Anatomic double-bundle ACL reconstruction will result in more symmetrical laxity and better range of motion and hop test scores in comparison to single-bundle ACL reconstruction.

Hypothesis 2.2 In comparison to single-bundle ACL reconstruction, anatomic double-bundle ACL reconstruction will result in better patient-oriented outcomes, indicating fewer symptoms, a higher level of activity and more complete return to sport.

Successful completion of these aims will provide quantitative evidence of the efficacy of anatomic double-bundle ACL reconstruction for restoring normal knee mechanics. Should the results show a clear benefit for this procedure, it would provide support for wider adaptation of anatomic DB reconstruction. By completing the proposed aims, we will also establish a sound basis for additional studies with longer follow-up (including the subjects in this cohort), to assess the benefits of anatomic DB ACL reconstruction for improving long-term clinical outcomes and maintaining joint and cartilage health.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) reconstruction is the 6th most common orthopaedic procedure. Disruption of the ACL leads to altered knee function and significantly increases the risk for osteoarthritis (OA). Current methods to reconstruct the ACL are generally perceived to be successful; however, several recent meta-analyses have indicated that normal structure and function of the knee is restored only 60% to 70% of the time and 60 to 90% have radiographic evidence of knee OA within 10 to 20 years. Though the causes of post-traumatic OA are almost certainly multifactorial, a significant factor contributing to the increased risk for OA following ACL injury and surgery may be failure to restore normal anatomy and kinematics of the knee.

We have previously shown that conventional single-bundle (SB) ACL reconstruction fails to restore normal knee kinematics, leading to altered patterns of joint loading. There is growing support for the theory that cartilage adapts to its local loading environment and abnormal joint loading may play an important role in the development and progression of OA. Our understanding of ACL anatomy has also improved over the last few years, revealing the shortcomings of current surgical techniques to restore anatomy of the ACL. We have developed double-bundle (DB) surgical procedures to restore normal anatomy of the anteromedial (AM) and posterolateral (PL) bundles of the ACL. The underlying principle for this approach is that more anatomical graft placement will lead to better knee mechanics, which are necessary for improved long-term outcome.

To determine if anatomic DB ACL reconstruction can effectively restore normal dynamic knee function, we will conduct a double-blind randomized clinical trial to compare SB vs. anatomic DB ACL reconstruction. The specific aims of this study are to determine if DB is better than SB ACL reconstruction in terms of 1) dynamic knee function and 2) clinical outcomes. We will randomly assign 160 subjects with an isolated ACL injury to SB or DB ACL reconstruction and will follow the subjects for 2 years. We will utilize a unique combination of high-speed biplane radiography (for accurate assessment of knee kinematics) and 3D imaging (MRI and CT, to define joint and cartilage morphology) to characterize joint kinematics and cartilage surface interactions during functional tasks. Clinical outcomes will include laxity, range of motion, functional strength and patient-reported symptoms, function and activity. Successful completion of this study will provide evidence of the efficacy of anatomic DB ACL reconstruction for restoring normal knee mechanics and improving clinical outcomes. If the results show a clear benefit of this procedure, then a sound basis will have been established for future studies to assess the benefits of anatomic DB ACL reconstruction on long-term clinical outcomes and joint health.

ELIGIBILITY:
Inclusion Criteria - subjects will be included in the study if they:

* Are between 14 and 50 years of age;
* Are scheduled for ACL reconstruction within 1 year of injury;
* Participate for greater than 100 hours per year in Level I (e.g. football, basketball or soccer) or Level II (e.g. racquet sports, skiing, manual labour occupations) activities;
* Have injury to both bundles of the ACL;
* Have tibial and femoral insertion sites that measure between 14 to 18 mm in diameter, as confirmed at the time of surgery;
* Have a femoral notch that is greater than or equal to 12 mm in width as measured with an arthroscopic ruler at the time of surgery and
* Are willing to continue participation in the study and return for all scheduled follow-up visits, even if he/she moves from the region.

Exclusion Criteria - Subjects will be excluded from participation in the study if they:

* Had prior surgery of the involved knee;
* Had a prior or currently have injury or surgery to the contra-lateral knee;
* Have open femoral or tibial growth plates as evidenced on the preoperative standard of care radiographs;
* Have greater than a grade I concomitant ligament injury;
* Have an Outerbridge grade 3 or 4 full thickness articular cartilage injury;
* Have evidence on the preoperative clinical MRI of insertional or intratendinous degeneration of the quadriceps tendon;
* Have a quadriceps tendon that is less than 7 mm thick on a sagittal cut of the preoperative clinical MRI;
* Have inflammatory or other forms of arthritis;
* Have any other injury or condition involving the lower extremity that affects the subjects' ability to walk or participate in Level I and II activities.

Because participation in this study requires subjects to undergo a research-related MRI, subjects will also be excluded if they:

* Had prior surgery for an aneurysm;
* Had any surgery within the past two months;
* Have a cardiac pacemaker;
* Have metal fragments in the eyes, brain or spinal cord;
* Have surgical implants;
* Have a history of claustrophobia or
* Have a history of not tolerating previous MRI scans without medication.

Women who are pregnant at the time of study enrollment or who plan to become pregnant within the 2 year follow-up period will not be eligible for participation in the study. If a female should become pregnant during the course of follow-up, kinematic testing, which would expose the fetus to radiation would be suspended until the pregnancy is complete.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2011-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Side to side difference in peak stance phase knee adduction | 6 months
  This is one of three primary outcomes for hypothesis 1.1 which states that knee kinematics after anatomic double-bundle ACL reconstruction are more similar to the uninjured contra-lateral limb than after single-bundle ACL reconstruction, as measured with dynamic stereoradiography 6 months after surgery. The side to side difference in peak stance-phase knee adduction was chosen because previous studies have shown that this variable was one that was most different from normal after single-bundle ACL reconstruction.
Side to side difference in peak stance-phase knee external rotation | 6 months
  This is one of three primary outcomes for hypothesis 1.1 which states that knee kinematics after anatomic double-bundle ACL reconstruction are more similar to the uninjured contra-lateral limb than after single-bundle ACL reconstruction, as measured with dynamic stereoradiography 6 months after surgery. The side to side difference in peak stance-phase knee external rotation was chosen because previous studies have shown that this variable was one that was most different from normal after single-bundle ACL reconstruction.
Side to side difference in peak stance-phase anterior tibial translation | 6 months
  This is one of three primary outcomes for hypothesis 1.1 which states that knee kinematics after anatomic double-bundle ACL reconstruction are more similar to the uninjured contra-lateral limb than after single-bundle ACL reconstruction, as measured with dynamic stereoradiography 6 months after surgery. The side to side difference in peak stance-phase anterior tibial translation was chosen because it is assumed that one of the primary functions of the ACL is to limit anterior tibial translation.
Relative change in graft elongation from 6 to 24 months | Difference from 6 to 24 months
  This is the primary outcome for hypothesis 1.2. Peak stance phase functional graft length will be measured 6 and 24 months after surgery with dynamic stereoradiography during walking and downhill running. For those that underwent double-bundle ACL reconstruction, functional graft length will be determined for both the anteromedial and posterolateral bundles. The relative change in graft elongation will be defined as the increase in peak functional graft length from 6 to 24 months normalized to functional graft length at 6 months.
Pivot shift test | 24 months
  This is 1 of 2 primary outcomes for hypothesis 2.1, which states that anatomic double-bundle ACL reconstruction will result in more symmetrical laxity and better range of motion and hop test scores in comparison to single-bundle ACL reconstruction 24 months after surgery. The 4-level scale for the pivot shift test will be collapsed to a binary outcome - "normal" vs. "not normal" (nearly normal, abnormal or severely abnormal).
Side to side difference in 30 lb. KT-1000 knee ligament arthrometer | 24 months
  This is 1 of 2 primary outcomes for hypothesis 2.1, which states that anatomic double-bundle ACL reconstruction will result in more symmetrical laxity and better range of motion and hop test scores in comparison to single-bundle ACL reconstruction 24 months after surgery. The side to side difference for the 30 lb KT-1000 test will be calculated.
IKDC Subjective Knee Form Score | 24 months
  This is the primary outcome for hypothesis 2.2, which states anatomic double-bundle ACL reconstruction will result in better patient-oriented outcomes, indicating fewer symptoms, a higher level of activity and more complete return to sports 24 months after surgery. The IKDC Subjective Knee Form is a validated 18-item patient reported measure of symptoms, activity and sports participation for individuals with a variety of knee conditions including ACL injury.
Side to side difference in peak stance phase knee adduction | 24 months
  This is one of three primary outcomes for hypothesis 1.1 which states that knee kinematics after anatomic double-bundle ACL reconstruction are more similar to the uninjured contra-lateral limb than after single-bundle ACL reconstruction, as measured with dynamic stereoradiography 6 and 24 months after surgery. The side to side difference in peak stance-phase knee adduction was chosen because previous studies have shown that this variable was one that was most different from normal after single-bundle ACL reconstruction.
Side to side difference in peak stance-phase knee external rotation | 24 months
  This is one of three primary outcomes for hypothesis 1.1 which states that knee kinematics after anatomic double-bundle ACL reconstruction are more similar to the uninjured contra-lateral limb than after single-bundle ACL reconstruction, as measured with dynamic stereoradiography 6 and 24 months after surgery. The side to side difference in peak stance-phase knee external rotation was chosen because previous studies have shown that this variable was one that was most different from normal after single-bundle ACL reconstruction.
Side to side difference in peak stance-phase anterior tibial translation | 24 months
  This is one of three primary outcomes for hypothesis 1.1 which states that knee kinematics after anatomic double-bundle ACL reconstruction are more similar to the uninjured contra-lateral limb than after single-bundle ACL reconstruction, as measured with dynamic stereoradiography 6 and 24 months after surgery. The side to side difference in peak stance-phase anterior tibial translation was chosen because it is assumed that one of the primary functions of the ACL is to limit anterior tibial translation.

SECONDARY OUTCOMES:
Joint contact path and velocity | 6 and 24 months
  This is a secondary outcome for hypothesis 1.1. The motion of the contact point in the medial and lateral compartments will be estimated during dynamic stereoradiography using MRI and CT scans to map bone and cartilage. The location of the centroid of the regions of cartilage overlap for the medial and lateral tibia and femur will be determined for each motion frame. The average velocity of the contact point along this path will be calculated for each bone surface.
Cartilage deformation and strain | 6 and 24 months
  This is a secondary outcome for hypothesis 1.1. Cartilage deformation and strain will be estimated as the area of cartilage overlap at the points of contact of the opposing bone surfaces in the medial and lateral compartment of the knee during walking and downhill running.
Side to side difference in knee range of motion | 3, 6, 12 & 24 months
  Side to side difference in knee range of motion is a secondary outcome for hypothesis 2.1. Passive extension and flexion of both knees will be measured with a goniometer and the side to side difference for each motion and well as for total motion of the knee will be calculated.
Hop tests | 6, 12 & 24 months
  The hop tests are a secondary outcome for hypothesis 2.1. The hop tests include 1) single leg hop for distance; 2) triple hop for distance; 3) triple cross over hop & 4) timed 10 m hop. Each of the tests will be performed on the contra-lateral normal and involved legs. For each of the tests, the involved leg will be expressed as a percentage of the non-involved leg and the average of the 4 hop tests will be calculated to represent the overall limb symmetry index.
Activities of Daily Living Scale of the Knee Outcome Score | 3, 6, 12, 24 months
  The Activities of Daily Living Scale (ADLS) of the Knee Outcome Score is a secondary outcome for hypothesis 2.2. The ADLS is a 14-item patient-reported measure of symptoms and activity limitations that was developed for individuals with a variety of knee impairments.
Knee injury and Osteoarthritis Outcomes Score | 3, 6, 1 & 24 months
  The Knee injury and Osteoarthritis Outcomes Score (KOOS) is a secondary outcome measure for hypothesis 2.2. The KOOS is a 42-item patient-reported outcome measure that results in 5 scores - pain, other symptoms, activities of daily living, sports & recreation and knee-related quality of life.
Veteran's RAND 12 Item Health Survey | 3, 6, 12 & 24 months
  The Veteran's RAND 12 Item Health Survey (VR-12) is a secondary outcome for hypothesis 2.2. The VR-12 was historically adapted from the SF-12 and results in physical and mental component summary scores that are standardized to the US population and norm based with a population mean of 50 and standard deviation of 10. The VR-12 was included because the scores can be converted to utilities that can be used for future evaluation of cost-effectiveness of single- vs. double-bundle ACL reconstruction.
Activity Measure for Post-Acute Care | 3, 6, 12 & 24 months
  The Activity Measure for Post-Acute Care (AM-PAC) is a secondary outcome for hypothesis 2.2. The AM-PAC is a computer adaptive test that incorporates the use of item response theory to measure basic mobility, daily activity and applied cognitive function. For this study, we will use the AM-PAC to measure only basic mobility.
Cincinnati Occupational Rating Scale | 3, 6, 12 & 24 months
  The Cincinnati Occupational Rating Scale is a secondary outcome for hypothesis 2.2. The Cincinnati Occupational Rating Scale is an 8-item measure of customary work activity. To complete this measure, subjects rate the frequency or duration of sitting, standing and walking, walking on uneven ground, squatting, climbing, lifting and carrying as well as the amount of weight that they routinely carry while at work.
Marx Sports Activity Scale | 3, 6, 12 & 24 months
  The Marx Sports Activity Scale is a secondary outcome for hypothesis 2.2. The Marx Sports Activity Scale is a 4-item patient-reported measure of sports activity. To complete the Marx Sports Activity Scale, subjects rate the frequency of performance of running, cutting, decelerating and pivoting.

CONTACTS AND LOCATIONS:
Overall Officials: James J Irrgang, PT PhD ATC, Principal Investigator — University of Pittsburgh; Freddie H Fu, MD, Principal Investigator — University of Pittsburgh; Scott Tashman, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Center for Sports Medicine, Pittsburgh, Pennsylvania, United States